CLINICAL TRIAL: NCT05572970
Title: Expanded Access for Cancer Treatment With Balstilimab (AGEN2034), Either as Monotherapy, or as Used in Combination With Zalifrelimab (AGEN1884)
Brief Title: Expanded Access for Cancer Treatment With Balstilimab (AGEN2034) and Zalifrelimab (AGEN1884)
Status: Available | Type: Expanded Access
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C-750-EAP-01
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: Balstilimab; AGEN2034; Zalifrelimab; AGEN1884; Monotherapy
MeSH Terms: conditions — Neoplasms | interventions — balstilimab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Balstilimab — An anti-programmed death 1 (PD-1) monoclonal antibody.
  Other Names: AGEN2034
Drug: Zalifrelimab — An anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) monoclonal antibody.
  Other Names: AGEN1884

SUMMARY:
This is an expanded access study for cancer treatment with balstilimab alone or in combination with zalifrelimab for an intermediate-size participant population. This study addresses the treatment needs of participants who have been previously and specifically treated with balstilimab alone or in combination with zalifrelimab in a clinical study, who have experienced a benefit from this treatment and/or wish to continue treatment, and who are eligible for treatment under this expanded access study.

DETAILED DESCRIPTION:
This study will not exceed 100 participants. Participants will be reevaluated annually to assess the treatment benefit of zalifrelimab and/or balstilimab and thereby, continued eligibility for treatment. Under this program, treatment will be continued with balstilimab, as either monotherapy or as used in combination therapy with zalifrelimab, for participants that have previously received one or both of these investigational medicinal products in a clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed predicate study protocol requirements, including prior treatment duration and follow-up.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - Hoag Gynecologic Oncology, Newport Beach, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Texas Oncology, Flower Mound, Texas